CLINICAL TRIAL: NCT05024123
Title: Pharmacokinetic Effect of AstraGin on Arginine Absorption and Nitric Oxide Production in Healthy Subjects: A Randomized, Double-blind, Crossover Trial
Brief Title: Pharmacokinetic Effect of AstraGin on Arginine Absorption and Nitric Oxide Production in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CS2-20203
Record Dates: First submitted 2021-05-20; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Absorption of Amino Acids and Peptides
Keywords: AstraGin; arginine; pharmacokinetic; nitric oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Experimental (Experimental)
  Interventions: Dietary Supplement: AstraGin

INTERVENTIONS:
Dietary Supplement: Placebo — Before each study day, the participants were subjected to a reduced nitrate content diet (avoid foods such as dark chocolate, beets, garlic, nuts and seeds, bacon, ham, and hot dogs,, day-1) for 24h. All subjects took a 50 mg placebo (maltodextrin) capsule at 9 p.m. and began fasting for 12 hours, except for a small amount of water in the night before the experiment. On each study day, all subjects collected their first blood sample at 9 a.m. from the median cubital vein using the indwelling catheter method. After the first blood collection, all subjects took 50 mg placebo and 5 g of L-arginine with 250 mL water.
  Additional blood samples were collected at 0, 15, 30, 45, 60, 90, 120, 150, and 180 min for analysis of the plasma concentration of amino acids, total nitrite, nitrate, and asymmetric dimethylarginine (ADMA) content.
  All subjects collected their urine during 0 ~ 180 min to measure 1) nitrate and 2) cGMP content.
  Arms: Placebo
Dietary Supplement: AstraGin — Before each study day, the participants were subjected to a reduced nitrate content diet (avoid foods such as dark chocolate, beets, garlic, nuts and seeds, bacon, ham, and hot dogs,, day-1) for 24h. All subjects took a 50 mg placebo (maltodextrin) capsule at 9 p.m. and began fasting for 12 hours, except for a small amount of water in the night before the experiment. On each study day, all subjects collected their first blood sample at 9 a.m. from the median cubital vein using the indwelling catheter method. After the first blood collection, all subjects took 50 mg placebo and 5 g of L-arginine with 250 mL water.
  Additional blood samples were collected at 0, 15, 30, 45, 60, 90, 120, 150, and 180 min for analysis of the plasma concentration of amino acids, total nitrite, nitrate, and asymmetric dimethylarginine (ADMA) content.
  All subjects collected their urine during 0 ~ 180 min to measure 1) nitrate and 2) cGMP content.
  Arms: Experimental

SUMMARY:
AstraGin increases the absorption of amino acids and peptides in Caco-2 cells and in normal and TNBS-induced rats. Given the potential beneficial applications of AstraGin for health, the effects on L-arginine uptake and nitric oxide production are investigated. The study is the L-arginine pharmacokinetic study: A randomized, double-blind, crossover trial. This study performed in healthy human subjects. The knowledge gained from this study will provide valuable information for the development of novel and effective natural food supplements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults and age 20 years and above, subdivided into three groups, Early-life (younger than 45 years, midlife (45--65 years), and later-life (older than 65 years), respectively.
* Subject has provided written and dated informed consent to participate in the study.
* The subject is willing and able to comply with the study.

Exclusion Criteria:

* The subject is participating in another clinical trial thirty days prior to enroll-ment.
* Subject has diabetes, obesity, hypertension, cardiovascular disease, liver or kid-ney disease, current infections, and smoking were exclusion criteria.
* Subject has any medical condition or uses any medication, nutritional product, amino acids supplement or program which might interfere with the conduct of the study or place the subject at risk.
* Subjects lost to follow-up, non-compliance, concomitant medication.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 3 hours
  Pharmacokinetic ( 0, 15, 30, 45, 60, 90, 120, 150, and 180 minutes)
Maximum Time [Tmax] | 3 hours
  Pharmacokinetic ( 0, 15, 30, 45, 60, 90, 120, 150, and 180 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan